CLINICAL TRIAL: NCT04315116
Title: A Single Center, Single Arm, Open and Fixed Sequence Study to Investigate the Pharmacokinetic Effects of Loperamide on Pyrotinib Maleate in Healthy Subjects
Brief Title: A Drug-drug Interaction Trial of Loperamide Pharmacokinetics Effect on Pyrotinib Maleate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HR-BLTN-DDI-04
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2020-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Loperamide

STUDY DESIGN:
Intervention Model Description: single arm, open and fixed sequence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treament (Experimental): Subjects receiving a single oral dose of pyrotinib maleate and wash-out for 6 days, then receiving Loperamide 4 mg bid from day 7 to day 13, with a single oral dose of pyrotinib maleate coadministered on day 10 .
  Interventions: Drug: pyrotinib maleate; Drug: Loperamide

INTERVENTIONS:
Drug: pyrotinib maleate — a single oral dose of pyrotinib maleate on day 1 & day10 .
Drug: Loperamide — Loperamide 4 mg bid from day 7 to day 13

SUMMARY:
The primary objective of the study was to assess the effect of repeated oral doses of Loperamide on the pharmacokinetic profile of a single dose of Pyrotinib Maleate.

The secondary objective of the study was to assess the safety of Pyrotinib Maleate given alone versus Fluzoparib coadministered with Loperamide.

ELIGIBILITY:
Inclusion Criteria:

* 1) Sign the informed consent form before the trial and fully understand the trial content, process and possible adverse reactions; 2) Ability to complete the study as required by the protocol; 3) Age on the date of signing the informed consent form is 18 to 45 years old (including both ends); 4) The fasting weight is not less than 50kg (male) and 45kg (female), and the body mass index (BMI) is in the range of 19 kg/m2 to 26 kg/m2 (including both ends);

Exclusion Criteria:

* 1) Participate in blood donation within 3 months before screening and donate blood volume ≥400mL or blood loss ≥400mL, or receive blood transfusion; 2) Allergic constitution, including a history of severe drug allergy or drug allergy; a history of allergies to Pyrotinib/ Loperamide capsule or its excipients; 3) with drug and/or alcohol abuse history, or alcohol and drug screening positives, or drug abuse in the past five years or used drugs 3 months before the trial; 4) Patients with bad habits (such as drinking 14 units of alcohol per week: 1 unit = 285mL of beer, 25mL of spirits, or 100mL of wine), smoking addiction (≥5 cigarettes per day);and could not prohibit smoking and alcohol during the trial period ; 5) QTc interval ≥ 450 ms in males and ≥ 470 ms in females; 6) left ventricular ejection fraction (LVEF) < 50% by echocardiography; 7) Other important organ diseases such as the nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolic and musculoskeletal system with clear medical history (such as uncontrolled diabetes, high blood pressure, etc.), enabling investigators considered unsuitable for participation in the study; 8) Anyone who has undergone any surgery within the first 6 months of screening; 9) Take any hepatotoxic drugs (eg dapsone, erythromycin, fluconazole, ketoconazole, rifampicin, etc.) within the first 6 months of screening; 10) Those who have taken any clinical trial drugs within 3 months; 11) Take any drug that affects liver metabolism within 4 weeks before taking the investigational drug; 12) Take any prescription or over-the-counter medication, vitamin products or herbs within 2 weeks before taking the investigational drug; 13) Clinical laboratory tests are abnormal and clinically significant, or other clinical findings indicate the following diseases, including but not limited to gastrointestinal, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular disease; 14) Female subjects during pregnancy, lactation, and subjects who were unable to abstain or take effective non-drug contraceptives during the study period and for at least 3 months after the last study drug administration (for female subjects Require abstinence or effective non-drug contraceptives two weeks before study entry); 15) combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive) or combined with syphilis infection; 16) Anyone who has ingested grapefruit or grapefruit-containing products, foods or drinks containing caffeine, xanthine or alcohol; strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion Within 48 hours; 17) Anyone who has pseudoulcerative colitis caused by acute ulcerative colitis or broad-spectrum antibiotics, or those who need to avoid inhibition of bowel movements, especially patients with intestinal obstruction, flatulence or constipation, or have diarrhea, dry mouth, Gastrointestinal symptoms such as bloating, loss of appetite, gastrointestinal cramps, nausea, vomiting, constipation, and dizziness, headache, and fatigue; 18) Anyone who has special requirements for diet and cannot comply with the diet and corresponding regulations provided by the test; 19) Anyone who has a history of dizzy needles and blood halo, who have difficulty collecting blood or cannot tolerate venipuncture; 20) The investigator believes that the subjects are not eligible to participate in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of pyrotinib | through study completion, an average of 20 days
  Peak Plasma Concentration (Cmax) of pyrotinib
Pharmacokinetics parameter: AUC of pyrotinib | through study completion, an average of 20 days
  Area under the plasma concentration versus time curve (AUC) of pyrotinib

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Tmax of pyrotinib | through study completion, an average of 20 days
  Time of maximum observed concentration (Tmax) of pyrotinib
Pharmacokinetics parameter: T1/2 of pyrotinib | through study completion, an average of 20 days
  Time of maximum observed concentration (Tmax) of pyrotinib
Pharmacokinetics parameter: CL/F of pyrotinib | through study completion, an average of 20 days
  Total body clearance for extravascular administration (CL/F) of pyrotinib
Pharmacokinetics parameter: Vz/F of pyrotinib | through study completion, an average of 20 days
  Volume of distribution (Vz/F) of pyrotinib
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion, an average of 20 days
  An adverse event is any untoward medical occurrence in a patient or clinical study participant

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No